CLINICAL TRIAL: NCT02985632
Title: Single-dose Pharmacokinetics of BMS-986141 in Participants With Hepatic Impairment Compared to Healthy Participants
Brief Title: A Study to Evaluate the Pharmacokinetics of BMS-986141 in Participants With Hepatic Impairment Compared to Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV006-030
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — BMS-986141

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild Hepatic Impairment Subjects (Experimental): Subjects given an oral dose of BMS-986141.
  Interventions: Drug: BMS-986141
- Moderate Hepatic Impairment Subjects (Experimental): Subjects given an oral dose of BMS-986141.
  Interventions: Drug: BMS-986141
- Healthy Subjects (Experimental): Subjects given an oral dose of BMS-986141.
  Interventions: Drug: BMS-986141

INTERVENTIONS:
Drug: BMS-986141

SUMMARY:
An oral dose of BMS-986141 administered in Hepatic Impairment and Healthy Participants to evaluate pharmacokinetics in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Women not of childbearing potential (WNOCBP), and males, ages 18 to 70 years, inclusive.
* BMI of 20.0 to 38.0 kg/m2 inclusive
* Participants who a history of normal renal function
* Subjects with hepatic impairment must be on a stable dose of medication and/or treatment regimen
* Healthy subjects to the extent possible matched to four subjects with hepatic impairment with regard to body weight, age and gender, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Any nonhepatic significant acute or chronic medical illness that could affect participant safety or data interpretation as determined by the investigator.
* History of recurrent dizziness or fall risk within 4 weeks of study drug administration
* History of primarily cholestatic liver diseases, autoimmune liver disease, metastatic liver disease or active alcoholic hepatitis
* History of known bleeding diathesis or coagulation disorder (eg, thrombotic thrombocytopenic purpura)
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-11 (Estimated); Primary Completion 2017-05-18 (Estimated); Study Completion 2017-07-07 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986141 | Days 1-7 (healthy) Days 1-10 (heaptic Impairment)
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-986141 | Days 1-7 (healthy) Days 1-10 (heaptic Impairment)
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of BMS-986141 | Days 1-7 (healthy) Days 1-10 (heaptic Impairment)
Area under the plasma concentration-time curve from time zero to 144 hours postdose (AUC(0-144h)) of BMS-986141 | Days 1-7 (healthy) Days 1-10 (heaptic Impairment)

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), leading to discontinuation. | Days 1-7 (healthy) Days 1-10 (heaptic Impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/